CLINICAL TRIAL: NCT07072624
Title: Assessing Phenytoin and Levetiracetam Efficacy, Cost-Effectiveness, and CYP2C9/SV2A Polymorphism in Early Post-Traumatic Seizures: A Multicentric Prospective Randomized Trial
Brief Title: Early Post-Traumatic Seizures Prevention Trial (E-PTS Trial)
Acronym: E-PTS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Jodhpur (Other Government)
Collaborators: Indian Council of Medical Research (Other Government); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Sanjay Gandhi Postgraduate Institute of Medical Sciences,Lucknow (Unknown)
Responsible Party: Principal Investigator, Jaskaran Singh Gosal, Associate Professor, All India Institute of Medical Sciences, Jodhpur
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIIMS/IEC/2024/4889; IIRPIG-2023-0001210 (Other Grant/Funding Number: Indian Council of Medical Research, Delhi)
Record Dates: First submitted 2025-05-30; First posted 2025-07-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Seizures; Traumatic Brain Injuries; Traumatic Brain Injury (TBI) Patients
Keywords: Post Traumatic Seizures; Early Post Traumatic Seizures; Traumatic Brain Injury; Seizure Prophylaxis; Antiepileptic drugs; Phenytoin; Levetiracetam; Placebo; Genetic polymorphism; CYP2C9; SV2A; Randomized Controlled Trial; Cost-effectiveness; Multicentric Trial
MeSH Terms: conditions — Seizures; Brain Injuries, Traumatic; Epilepsy, Post-Traumatic | interventions — Phenytoin; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phenytoin (Active Comparator)
  Interventions: Drug: Phenytoin
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenytoin — The Phenytoin group will be given a loading dose of phenytoin 20 mg/kg intravenously (maximum, 2 gm) at 50 mg per minute and then started on a maintenance dose (5-6 mg/kg/d, rounded to the nearest 100 mg, intravenously administered every 8 hours). The intravenous will be switched to oral once the patient is fit to take it orally or via Ryles tube. The oral dose would be a single 300 mg ER (extended-release) tablet per day. Both IV and/or oral doses of phenytoin will be given only for 1 week after head trauma. Patient= Patients with Traumatic brain injury as per eligibility criteria. Intervention= Phenytoin loading dose IV (20 mg/kg) followed by 100 mg IV TDS till patient accepts orally. Oral dose will be administered as a single 300 mg ER tablet per day. Both IV and oral phenytoin will be given for 1 week after traumatic brain injury and then stopped. Comparator= Matching Placebo
  Arms: Phenytoin
Drug: Levetiracetam — The Levetiracetam group will receive 25-30 mg/kg/d in two divided doses (rounded to 750 mg, administered intravenously every 12 hourly). The intravenous dose will be switched to oral form once the patient is fit to take it orally or via Ryles tube. The oral dose would be two tablets of 750 mg ER (extended-release) levetiracetam daily. Both IV and/or oral doses of levetiracetam will be given only for 1 week after head trauma. Patient= Patients with Traumatic brain injury as per eligibility criteria. Intervention= Levetiracetam IV dosing will be 25-30 mg/Kg/d in 2 divided doses (rounded to 750 mg IV BD) followed by 2 tablets of 750 mg ER once patient fit to take orally or via Ryles tube. Comparator= Matching Placebo.
  Arms: Levetiracetam
Drug: Placebo — The Placebo group will be administered normal saline intravenously of similar amount that of intervention group and matching placebo tablets orally (double dummy) once the patient is fit to take orally. Similar to the intervention group, both IV and oral placebo will be given till 1 week after traumatic brain injury.
  Arms: Placebo

SUMMARY:
Rationale/gaps in existing knowledge: The prophylaxis for post-traumatic seizures (PTS) remains controversial due to a lack of class I evidence. Investigators plan to conduct a high-quality, prospective, multicentric, randomized study regarding seizure prophylaxis in traumatic brain injury (TBI) with phenytoin, levetiracetam, and the placebo in three respective treatment groups, along with the effect of drug polymorphism on seizure occurrence.

Novelty: Literature is scarce regarding the ideal management of early PTS in traumatic brain injury (TBI), a major public health problem. Further, no study has evaluated the effect of genetic polymorphism on seizure occurrence in traumatic brain injury. This Multicentric study will be the first of its kind, not only in India but also globally.

Objectives: To evaluate the seizure incidence & efficacy of the respective anti-epileptic drug in each treatment arm. Assessment of clinical & functional outcomes, safety profile, and cost-effectiveness in each group. Effect of genetic polymorphisms on seizure incidence among study participants Methods: A Multicentric prospective randomized placebo-controlled double-blinded clinical trial is planned. After satisfying eligibility criteria and informed consent, TBI patients will be randomly allocated into three arms 'phenytoin arm', 'levetiracetam arm', and 'placebo'. Drug polymorphism will be analyzed in all the patients using quantitative real-time PCR.

Expected outcome: This study will provide high-quality evidence in PTS management and will establish the role of prophylactic anti-epileptics in PTS. This study also opens the plethora of undesignated roles of genetic polymorphism in the efficacy and safety of levetiracetam and phenytoin in traumatic brain injury patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of severe blunt TBI with GCS score less than 10.
2. Patients with GCS of more than 10 in the presence of computed tomographic imaging findings consistent with brain injury: subarachnoid hemorrhage [SAH], subdural hematoma [SDH], epidural hematoma [EDH], intracerebral hemorrhage [ICH], or diffuse axonal injury [DAI], depressed skull fracture.
3. Patients with penetrating injury.

Exclusion Criteria:

1. Females of childbearing age with urine pregnancy test positive.
2. Devastating brain injury with expected or confirmed brain death within 48 hours of hospital admission,
3. Prehospital use of anticonvulsants
4. Development of seizures before enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Clinical Seizure Within 7 Days Post-Traumatic Brain Injury in each of the three treatment groups. | 7 Days
  A total of 1260 participants experiencing early clinical seizures (defined as any observable seizure activity occurring within 7 days post-trauma), as recorded by treating clinicians, and confirmed through clinical documentation, during the first 7 days of the study intervention period in each group (Phenytoin, Levetiracetam, Placebo).

SECONDARY OUTCOMES:
Change in Glasgow Coma Scale scores from baseline at 7 days post-trauma, at 6 months, and 1 year in each treatment group. | 7 Days , 6 Months & 1 year
  Title: Functional and Neurological Status Assessed Using Glasgow Coma Scale (GCS).
  Description:
  Glasgow Coma Scale (GCS)-a clinical tool used to assess the level of consciousness in traumatic brain injury patients. Scores range from 3 to 15, where higher scores indicate better neurological function. The GCS differentiates between the severities of head injury by score ranges. A GCS of 13-15 indicates a mild head injury, 9-12 moderate and 3-8 severe.
  Time Frame:
  GCS: Day 1(Baseline), Day 3, Day 5, and Day 7, at discharge , at 6-month & 1 year follow up.
  Assessment Method:
  GCS: Assessed by trained clinical staff daily using standard scoring protocol.
Glasgow Outcome Scale scores at hospital discharge, 6-month, and 1-year follow-up in each treatment group. | At discharge, 6 months and 1 year
  Title: Functional and Neurological Status Assessed Using Glasgow Outcome Scale (GOS).
  Description: Glasgow Outcome Scale (GOS) - a global outcome measure of functional recovery post-TBI. Scores range from 1 (death) to 5 (good recovery), where higher scores indicate better outcomes.
  Time Frame: GOS: At hospital discharge and 6-month follow-up. Assessment method GOS: Assessed at discharge by clinical staff, and at 6 months and at 1 year via telephonic or in-person follow-up
Incidence of early clinical seizures in participants, assessed in association with CYP2C9 and SV2A gene polymorphisms, using TaqMan allelic discrimination assay with quantitative real-time PCR (qPCR). | 7 days
  Title:
  Association Between CYP2C9 and SV2A Genetic Polymorphisms and Early Seizure Incidence.
  Description: Genotyping of CYP2C9 and SV2A polymorphisms will be performed using TaqMan allelic discrimination assay with quantitative real-time PCR. The incidence of early clinical seizures (defined as seizures occurring within 7 days post-trauma) will be compared across different genotype groups. The outcome will be reported as the number and proportion of participants with early seizures by genotype.
  Time Frame: Within 7 days post-injury Unit of Measure: Number of participants with seizures per genotype group.
Incremental Cost-Effectiveness Ratio (ICER) of Levetiracetam vs Phenytoin in Preventing Early Post-Traumatic Seizures using Markov chain Monte Carlo simulation. | 1 year
  Description: Cost-effectiveness within the trial will be assessed by calculating the Incremental Cost-Effectiveness Ratio (ICER), defined as the difference in direct medical costs per seizure complication prevented between the phenytoin and levetiracetam groups.
  Cost data include direct medical cost like drug acquisition, hospital stay, ICU stay, investigations, and seizure-related interventions. Outcome data will include the number of patients with early clinical seizures (within 7 days).
  Economic evaluation will be performed over a 1-year follow-up period using trial-based data. ICER values will be calculated along with 95% confidence intervals, and sensitivity analyses will be conducted using probabilistic approach. Long-term cost effectiveness will be modelled using Markov chain Monte Carlo simulation.
  Time Frame: From randomization to 1-year post-injury follow-up. Measure Type: Cost-effectiveness ratio Unit of Measure: INR (₹) per seizure prevented

CONTACTS AND LOCATIONS:
Overall Officials: Dr Apinderpreet Singh Additional Professor, MCh Neurosugery, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Dr Kamlesh Bhaisora Additional Professor, MCh Neurosugery, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences,Lucknow
Locations (3):
- India (3):
  - Postgraduate Institute of Medical Education & Research, Chandigarh, Punjab
  - AIIMS Jodhpur, Jodhpur, Rajasthan
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta V, Gupta K, Singh G, Kaushal S. An Analytical Study to Correlate Serum Levels of Levetiracetam with Clinical Course in Patients with Epilepsy. J Neurosci Rural Pract. 2016 Dec;7(Suppl 1):S31-S36. doi: 10.4103/0976-3147.196445. PMID 28163500
- [Background] Kousar S, Wafai ZA, Wani MA, Jan TR, Andrabi KI. Clinical relevance of genetic polymorphism in CYP2C9 gene to pharmacodynamics and pharmacokinetics of phenytoin in epileptic patients: validatory pharmacogenomic approach to pharmacovigilance. Int J Clin Pharmacol Ther. 2015 Jul;53(7):504-16. doi: 10.5414/CP202112. PMID 25943175
- [Background] Chang WC, Hung SI, Carleton BC, Chung WH. An update on CYP2C9 polymorphisms and phenytoin metabolism: implications for adverse effects. Expert Opin Drug Metab Toxicol. 2020 Aug;16(8):723-734. doi: 10.1080/17425255.2020.1780209. Epub 2020 Jul 16. PMID 32510242
- [Background] Dibbens LM, Hodgson BL, Helbig KL, Oliver KL, Mulley JC, Berkovic SF, Scheffer IE. Rare protein sequence variation in SV2A gene does not affect response to levetiracetam. Epilepsy Res. 2012 Sep;101(3):277-9. doi: 10.1016/j.eplepsyres.2012.04.007. Epub 2012 Apr 30. PMID 22551666
- [Background] Schivell AE, Mochida S, Kensel-Hammes P, Custer KL, Bajjalieh SM. SV2A and SV2C contain a unique synaptotagmin-binding site. Mol Cell Neurosci. 2005 May;29(1):56-64. doi: 10.1016/j.mcn.2004.12.011. PMID 15866046
- [Background] Jones KE, Puccio AM, Harshman KJ, Falcione B, Benedict N, Jankowitz BT, Stippler M, Fischer M, Sauber-Schatz EK, Fabio A, Darby JM, Okonkwo DO. Levetiracetam versus phenytoin for seizure prophylaxis in severe traumatic brain injury. Neurosurg Focus. 2008 Oct;25(4):E3. doi: 10.3171/FOC.2008.25.10.E3. PMID 18828701
- [Background] Szaflarski JP, Sangha KS, Lindsell CJ, Shutter LA. Prospective, randomized, single-blinded comparative trial of intravenous levetiracetam versus phenytoin for seizure prophylaxis. Neurocrit Care. 2010 Apr;12(2):165-72. doi: 10.1007/s12028-009-9304-y. PMID 19898966
- [Background] Jarvie D, Mahmoud SH. Therapeutic Drug Monitoring of Levetiracetam in Select Populations. J Pharm Pharm Sci. 2018;21(1s):149s-176s. doi: 10.18433/jpps30081. PMID 30096051
- [Background] Cardona AF, Rojas L, Wills B, Bernal L, Ruiz-Patino A, Arrieta O, Hakim EJ, Hakim F, Mejia JA, Useche N, Bermudez S, Carranza H, Vargas C, Otero J, Mayor LC, Ortiz LD, Franco S, Ortiz C, Gil-Gil M, Balana C, Zatarain-Barron ZL. Efficacy and safety of Levetiracetam vs. other antiepileptic drugs in Hispanic patients with glioblastoma. J Neurooncol. 2018 Jan;136(2):363-371. doi: 10.1007/s11060-017-2660-0. Epub 2017 Nov 25. PMID 29177594
- [Background] Dikmen SS, Temkin NR, Miller B, Machamer J, Winn HR. Neurobehavioral effects of phenytoin prophylaxis of posttraumatic seizures. JAMA. 1991 Mar 13;265(10):1271-7. PMID 1995974
- [Background] Bhullar IS, Johnson D, Paul JP, Kerwin AJ, Tepas JJ 3rd, Frykberg ER. More harm than good: antiseizure prophylaxis after traumatic brain injury does not decrease seizure rates but may inhibit functional recovery. J Trauma Acute Care Surg. 2014 Jan;76(1):54-60; discussion 60-1. doi: 10.1097/TA.0b013e3182aafd15. PMID 24368357
- [Background] Young B, Rapp RP, Norton JA, Haack D, Tibbs PA, Bean JR. Failure of prophylactically administered phenytoin to prevent late posttraumatic seizures. J Neurosurg. 1983 Feb;58(2):236-41. doi: 10.3171/jns.1983.58.2.0236. PMID 6848681
- [Background] Ferguson PL, Smith GM, Wannamaker BB, Thurman DJ, Pickelsimer EE, Selassie AW. A population-based study of risk of epilepsy after hospitalization for traumatic brain injury. Epilepsia. 2010 May;51(5):891-8. doi: 10.1111/j.1528-1167.2009.02384.x. Epub 2009 Oct 20. PMID 19845734
- [Background] Annegers JF, Hauser WA, Coan SP, Rocca WA. A population-based study of seizures after traumatic brain injuries. N Engl J Med. 1998 Jan 1;338(1):20-4. doi: 10.1056/NEJM199801013380104. PMID 9414327
- [Background] Temkin NR, Dikmen SS, Wilensky AJ, Keihm J, Chabal S, Winn HR. A randomized, double-blind study of phenytoin for the prevention of post-traumatic seizures. N Engl J Med. 1990 Aug 23;323(8):497-502. doi: 10.1056/NEJM199008233230801. PMID 2115976
- [Background] Torbic H, Forni AA, Anger KE, Degrado JR, Greenwood BC. Use of antiepileptics for seizure prophylaxis after traumatic brain injury. Am J Health Syst Pharm. 2013 May 1;70(9):759-66. doi: 10.2146/ajhp120203. PMID 23592358
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Inaba K, Menaker J, Branco BC, Gooch J, Okoye OT, Herrold J, Scalea TM, Dubose J, Demetriades D. A prospective multicenter comparison of levetiracetam versus phenytoin for early posttraumatic seizure prophylaxis. J Trauma Acute Care Surg. 2013 Mar;74(3):766-71; discussion 771-3. doi: 10.1097/TA.0b013e3182826e84. PMID 23425733
- [Background] Agrawal A, Munivenkatappa A, Shukla DP, Menon GR, Alogolu R, Galwankar S, Kumar SS, Momhan PR, Pal R, Rustagi N. Traumatic brain injury related research in India: An overview of published literature. Int J Crit Illn Inj Sci. 2016 Apr-Jun;6(2):65-9. doi: 10.4103/2229-5151.183025. PMID 27308253
- [Background] Gururaj G. Epidemiology of traumatic brain injuries: Indian scenario. Neurol Res. 2002 Jan;24(1):24-8. doi: 10.1179/016164102101199503. PMID 11783750
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556